CLINICAL TRIAL: NCT04445142
Title: Severe Foveal Epiretinal Membrane Contraction After Previous Fovea-sparing Internal Limiting Membrane Peeling Surgery
Brief Title: Fovea ERM After Fovea-sparing ILM Peeling
Status: Completed | Type: Observational
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, San Ni Chen, Head of department of ophthalmology, Changhua Christian Hospital
Other Study IDs: 200402
Record Dates: First submitted 2020-05-23; First posted 2020-06-24 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Epiretinal Membrane; Internal Limiting Membrane Wrinkling
Keywords: Fovea-sparing internal limiting membrane peeling; Epiretinal membrane.
MeSH Terms: conditions — Epiretinal Membrane

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- epiretinal membrane group: Patients developed secondary fovea epiretinal membrane
  Interventions: Procedure: fovea-sparing internal limiting membrane peeling

INTERVENTIONS:
Procedure: fovea-sparing internal limiting membrane peeling — fovea-sparing internal limiting membrane peeling surgery

SUMMARY:
To report cases who had received previous fovea-sparing internal limiting peeling membrane and developed secondary fovea epiretinal membrane contraction

DETAILED DESCRIPTION:
Purpose: To report the rare complication of foveal epiretinal membrane (ERM) formation on residual internal limiting membrane (ILM) with severe contraction after previous fovea-sparing internal limiting membrane (ILM) peeling.

Study design: Retrospective case series Methods: We report patients who previously received fovea-sparing ILM peeling and complicated with foveal ERM formation and contraction.

ELIGIBILITY:
Inclusion Criteria:

* patients who developed secondary fovea epiretinal membrane after previous fovea-sparing internal limiting membrane surgery

Exclusion Criteria:

* patients who did not receive previous fovea-sparing internal limiting membrane surgery

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients who developed secondary fovea epiretinal membrane after previous fovea-sparing internal limiting membrane surgery
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Visual acuity | 6 months
  Snellen visual acuity change
Optical coherence tomography finding | 6 months
  fovea change on optical coherence tomography

CONTACTS AND LOCATIONS:
Overall Officials: San-Ni Chen, MD, Study Chair — Changhua Christian Hospital
Locations (1):
- Department of ophthalmology, Changhua Christian Hospital, Changhua, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen YC, Chen SN. Isolated Central Epiretinal Membrane: A Rare Complication of Fovea-Sparing Internal Limiting Membrane Peeling Technique. J Ophthalmol. 2021 Apr 14;2021:6654604. doi: 10.1155/2021/6654604. eCollection 2021. PMID 33936809